CLINICAL TRIAL: NCT02250495
Title: VIBE: A Clinical Study to Evaluate the Sympara Therapeutic System for the Treatment of Hypertension
Brief Title: The Sympara VIBE Study for Hypertension
Acronym: VIBE
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company closed
Sponsor: Sympara Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STS1402
Record Dates: First submitted 2014-09-20; First posted 2014-09-26 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sympara Therapeutic System (Experimental): All subjects will wear for the Sympara device for 30 days
  Interventions: Device: Sympara Therapeutic System

INTERVENTIONS:
Device: Sympara Therapeutic System — Sympara Therapeutic System as a non-invasive, fully reversible alternative for the treatment of hypertension

SUMMARY:
The purpose of the VIBE study is to evaluate the efficacy and safety of the Sympara Therapeutic System in the treatment of hypertension

ELIGIBILITY:
Inclusion Criteria:

* Office systolic blood pressure of ≥150mmHg based on an average of three (3) blood pressure reading measured at both the initial screening visit and a confirmatory screening visit OR a mean daytime systolic blood pressure ≥135mm Hg on 24-hour Ambulatory Blood Pressure Measurement
* Receiving and adhering to an appropriate anti-hypertensive treatment regimen, as prescribed by physician
* Minimum six- (6) month history of diagnosis and treatment of hypertension

Exclusion Criteria:

* Previous renal denervation or carotid barostimulation implant
* Secondary causes of hypertension or primary pulmonary hypertension
* Prior surgery or radiation to the area of the carotid sinus, or presence of a stent or other implant in the carotid artery
* Known or suspected baroreflex failure or significant orthostatic hypotension
* One or more hospital admissions for a hypertensive crisis within the past year
* History of myocardial infarction, fibrillation event, unstable angina pectoris, syncope, transient ischemic attach (TIA) or a cerebrovascular accident within six (6) months of the screening period, or has widespread atherosclerosis with documented intrasvascular thrombosis or unstable plaques
* Diabetes mellitus (Type 1)
* Chronic renal disease requiring dialysis
* Kidney or liver transplant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with serious, device-related adverse events as a measure of safety and tolerability | 30 days

SECONDARY OUTCOMES:
Number of subjects with a reduction in baseline blood pressure following 30 days of Sympara device use as a measure of efficacy | 30 days
  Evaluating change in office, home and ambulatory blood pressure measurements at 30 days compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ian Meredith, AM, PhD, Principal Investigator — Monash Health
Locations (3):
- Australia (3):
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Monash Health, Clayton, Victoria
  - Barwon Health, Geelong, Victoria